CLINICAL TRIAL: NCT02974296
Title: Neuroimaging in Patients Undergoing TMS for Depression
Acronym: NIPUTFD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Marta Moreno Ortega, PHD, Associate Research Scientist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7159
Record Dates: First submitted 2016-11-18; First posted 2016-11-28 (Estimated); Results first posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- new target TMS (Experimental): new target transcranial magnetic stimulation guided by MRI
  Interventions: Device: transcranial magnetic stimulation
- standard TMS (Active Comparator): standard transcranial magnetic stimulation
  Interventions: Device: transcranial magnetic stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation — non invasive brain stimulation approach

SUMMARY:
The goal of this project is to guide rTMS using functional magnetic resonance imaging (fMRI) in individuals with depression who did not respond to standard TMS treatment to evaluate whether targeted TMS using individualized functional MRI scans produce outcome superior to that of conventional approaches. The study team also plans to scan patients with Major Depression Disorder (MDD) patients prescribed to receive standard TMS for the first time before and after which they will have resting-state Functional Magnetic Resonance Imaging (rs-FMRI) scan in order to see if we can predict their responsiveness based on the functional connectivity maps.

DETAILED DESCRIPTION:
Significance: There are few therapeutic options for individuals with treatment resistant depression (TRD). One recently developed approach is rTMS over left dorsolateral prefrontal cortex. Recent studies have demonstrated overall antidepressant benefit of rTMS in patients who fail to respond to a trial of antidepressant medication (1, 2, 3). Nevertheless, for many patients the response is incomplete, suggesting the need for further optimization. One potential cause of heterogeneous response might relate to individual differences in brain anatomy and connectivity patterns. At present, the rTMS stimulation site across subjects is based upon fixed location relative to motor cortex. Potentially, however, the approach could be optimized by stimulating based upon individual brain functional connectivity pattern. The present project will collect pre- and post-treatment brain functional connectivity measures in a group of patients who will be receiving independent clinical rTMS for resistant depression, a connectivity-based targeting approach will be applied at the single-subject level to individualize therapy in those patients who do not respond to standard approaches.

Patients will be divided in 2 groups. Group 1 (N=30) will be depressed patients undergoing standard TMS for the first time. Group 2 (N=30) constitutes those who have previously demonstrated that they do not respond to standard TMS. MDD patients prescribed to receive standard TMS for the first time (group 1) will have resting-state FMRI in order to see if their responsiveness based on the functional connectivity maps can be predicted. Non-responders to standard TMS approaches (Group 2) will be randomized (3:2) to either receive targeted (N=18) or standard (N=12) repetitive TMS (rTMS) treatments. A connectivity-based targeting strategy will be used on patients undergoing targeted rTMS to optimize target for focal brain stimulation. Raters and patients in group 2 will be kept blinded to the treatment assignment. All patients referred from the ongoing treatment study will be assessed by 3 tesla brain MRI, Magnetic Resonance Spectroscopy (MRS) and Cerebral Blood Flow/Volume (CBF/CBV) procedures at baseline and immediately following the final treatment.

ELIGIBILITY:
General Inclusion Criteria:

1. Male or female outpatients, 18 to 60 years of age.
2. Primary diagnosis of Major Depressive Disorder as confirmed by the Structured Clinical Interview for Diagnostic and Statistical Manual (DSM-IV-TR) Disorders (SCID-IV-TR).
3. Duration of the index episode of at least 1 month.
4. MDD symptoms, defined as a total HDRS-17 score ≥ 18 despite treatment with an adequate trial of a serotonin reuptake inhibitor (SRI).
5. Individuals who cannot tolerate medications.
6. Patients currently on medication must be at the same stable dose(s) for 1 month prior to enrollment and be willing to continue at the same dose(s) through the duration of the study.
7. Capable and willing to provide informed consent.
8. Signed HIPAA authorization.
9. Right-handed.
10. Willingness to undergo research fMRI scan (3T).
11. Willingness to undergo randomization to either treatment arm.

General Exclusion Criteria:

1. Investigators, and their immediate families (defined as a spouse, parent, child or sibling, whether by birth or legal adoption).
2. Individuals diagnosed by the investigators with the following conditions: Bipolar Disorder (lifetime), any Psychotic Disorder (lifetime), history of substance abuse or dependence within the past year (except nicotine and caffeine).
3. Behavior, which in the judgment of the investigator may hinder the patient in completing the procedures required by the study protocol.
4. Individuals with a clinically defined neurological disorder including, but not limited to: tics, space occupying brain lesion; any history of seizures except those therapeutically induced by electroconvulsive therapy (ECT); history of cerebrovascular accident; history of fainting; transient ischemic attack within two years; cerebral aneurysm, Dementia; Parkinson's Disease; Huntington chorea; Multiple Sclerosis.
5. Increased risk of seizure for any reason, including prior diagnosis of increased intracranial pressure (such as after large infarctions or trauma), or history of significant head trauma with loss of consciousness for ≥ 5 minutes.
6. Use of any investigational drug within 12 weeks of the randomization visit.
7. Significant acute suicide risk, defined as follow: suicide attempt within the previous 6 months that required medical treatment; or ≥ 2 suicide attempts in the past 12 months; or in the investigator's opinion, has significant risk for suicide based on the current state or recent history.
8. Cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease.
9. Intracranial implants (e.g. aneurysms clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed.
10. Current illicit drug use (cannabinoid, phencyclidine, amphetamines, barbiturates, cocaine, methadone, and opiates), defined as drug use during the 6 months before screening.
11. Known or suspected pregnancy. Urine pregnancy test Women who are breast-feeding.
12. Women of childbearing potential not using a medically accepted form of contraception when engaging in sexual intercourse.
13. Medicinal patch, unless removed prior to the magnetic resonance (MR) scan.
14. MDD patients with very severe depression, defined as a total HDRS-17 score ≥ 23, will be excluded and referred to immediate treatment.
15. Risks related to seizures, such as substance abuse or sleep disruptions/insomnia.

SpecificExclusion criteria (group 1):

History of treatment with rTMS therapy for any disorder.

Specific Inclusion criteria (group 2):

History of non-response to rTMS in this depressive episode.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2017-04-30 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C. Javitt, MD Ph.D, Study Director — New York State Psychiatric Institute & Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moreno-Ortega M, Kangarlu A, Lee S, Perera T, Kangarlu J, Palomo T, Glasser MF, Javitt DC. Parcel-guided rTMS for depression. Transl Psychiatry. 2020 Aug 12;10(1):283. doi: 10.1038/s41398-020-00970-8. PMID 32788580

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | New Target TMS | Standard TMS
Started | 10 | 23
Completed | 10 | 22
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | New Target TMS | Standard TMS | Total
Number analyzed (Participants) | 10 | 22 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 22 | 32
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.70 (16.028) | 41.50 (15.152) | 40.21 (15.275)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 12 | 15
  Male | 7 | 10 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 9 | 21 | 30
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 22 | 32

OUTCOME MEASURES:

1. Primary Outcome: Change in Functional Connectivity Measured by Resting MRI
Description: Change from Baseline in Resting MRI Correlation Coefficients Between Left Dorsolateral Prefrontal Cortex and Subgenual Anterior Cingulate Change in Resting MRI is defined as post-pre
Time Frame: Week 1 prior to first TMS treatment and week 36 after completion of TMS treatments
Measure: Mean (Standard Deviation); unit: correlation coefficients
Arm/Group | New Target TMS | Standard TMS
Number analyzed (Participants) | 10 | 22
correlation coefficients | 0.103399365 (0.161565183) | -0.7637409 (0.106948404)

2. Secondary Outcome: Change in Depressive Symptoms Measured by the Hamilton Depression Rating Scale (17-item HDRS)
Description: Patients will be classified as responders to TMS with at least 50% decrease in HDRS scores from baseline. Patients will be classified as non-responders to TMS with less than 50% decrease in HDRS scores from baseline.
  Change in HDRS-17 scores is defined as: [pre-post)/pre]x100 HDRS-17 scores range: 0-61
  Levels of depression based on HDRS-17 scores:
  Not depressed: 0-7 Mild (subthreshold): 8-13 Moderate (mild): 14-18 Severe (moderate): 19-22 Very severe (severe): >23
Time Frame: Week 1 prior to first TMS treatment and week 36 after completion of TMS treatments
Measure: Mean (Standard Deviation); unit: percentage change in HDRS scores
Arm/Group | New Target TMS | Standard TMS
Number analyzed (Participants) | 10 | 22
percentage change in HDRS scores | 64.9440 (15.16426) | 27.7345 (27.48549)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | New Target TMS | Standard TMS
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/22
Other Adverse Events (participants affected / at risk) | 0/10 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/96/NCT02974296/Prot_ICF_002.pdf
  • Statistical Analysis Plan (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/96/NCT02974296/SAP_003.pdf